CLINICAL TRIAL: NCT06910761
Title: Phase II Trial of Photon Craniospinal Irradiation for Leptomeningeal Disease Secondary to Solid Tumor Malignancy
Brief Title: Photon Craniospinal Irradiation for the Treatment of Leptomeningeal Disease Secondary to Breast Cancer or Non-small Cell Lung Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23911; NCI-2025-02015 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 23911 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2025-03-28; First posted 2025-04-04 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Anatomic Stage IV Breast Cancer AJCC v8; Metastatic Breast Carcinoma; Metastatic Lung Non-Small Cell Carcinoma; Metastatic Malignant Neoplasm in the Leptomeninges; Stage IV Lung Cancer AJCC v8
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Non-Small-Cell Lung; Meningeal Carcinomatosis; Lung Neoplasms | interventions — Specimen Handling; Craniospinal Irradiation; Spinal Puncture; Magnetic Resonance Spectroscopy; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Photon-VMAT-CSI) (Experimental): Patients undergo photon-VMAT-CSI QD for 10 treatments over 10-20 days (Monday-Friday) in the absence of disease progression or unacceptable toxicity. Patients undergo MRI during screening and follow-up and undergo collection of blood samples throughout the trial. Patients also undergo LP or Ommaya reservoir tap for CSF sample collection during screening and follow-up.
  Interventions: Procedure: Biospecimen Collection; Radiation: Craniospinal Irradiation; Other: Electronic Health Record Review; Procedure: Lumbar Puncture; Procedure: Magnetic Resonance Imaging; Procedure: Ommaya Reservoir Tap; Other: Questionnaire Administration; Radiation: Volume Modulated Arc Therapy

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood and CSF sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Radiation: Craniospinal Irradiation — Undergo photon-VMAT-CSI
Other: Electronic Health Record Review — Ancillary studies
Procedure: Lumbar Puncture — Undergo LP
  Other Names: LP; Spinal Tap
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Procedure: Ommaya Reservoir Tap — Undergo Ommaya reservoir tap
  Other Names: Ommaya Reservoir Access
Other: Questionnaire Administration — Ancillary studies
Radiation: Volume Modulated Arc Therapy — Undergo photon-VMAT-CSI
  Other Names: VMAT; Volumetric Modulated Arc Therapy (procedure)

SUMMARY:
This phase II trial tests how well craniospinal irradiation (CSI) using photon volumetric modulated arc radiotherapy (VMAT) works in treating patients with breast cancer or non-small cell lung cancer (NSCLC) that has spread from the original (primary) tumor to the cerebrospinal fluid and meninges (thin layers of tissue that cover and protect the brain and spinal cord) (leptomeningeal disease). Radiation therapy uses high energy x-rays, particles, or radioactive seeds to kill cancer cells and shrink tumors. CSI (radiation therapy directed at the brain and spinal cord to kill tumor cells) may be able to target all of the areas of possible leptomeningeal tumor spread. Photon-VMAT-CSI may be an effective treatment option for patients with leptomeningeal disease secondary to breast cancer or NSCLC.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the efficacy of photon-VMAT-CSI; assessed by median central nervous system progression free survival (CNS-PFS).

SECONDARY OBJECTIVES:

I. To estimate and assess central nervous system (CNS) response rate, response duration, and overall survival probability.

II. To summarize and assess toxicities including: type, frequency, severity, attribution, time course and duration.

III. To characterize and evaluate patient reported outcomes (PROs), including quality of life (QOL), measures:

IIIa. QOL Questionnaire Brain 20 (European Organization for Research and Treatment of Cancer [EORTC]-Quality of Life Questionnaire [QLQ]-Brain 20 [BN20]); IIIb. Core QOL Questionnaire 30 (EORTC-QLQ-Core 30 [C30]); IIIc. Patient reported outcomes measurement information system (PROMIS) for Anxiety; IIId. PROMIS Cognition.

EXPLORATORY OBJECTIVES:

I. To characterize inflammatory markers over time. II. To explore the potential association between inflammatory markers and radiation-related toxicity.

III. To evaluate the potential association between circulating cell-free deoxyribonucleic acid (cfDNA), imaging, and response.

IV. To evaluate possible genomic predictors of CNS progression.

OUTLINE:

Patients undergo photon-VMAT-CSI once daily (QD) for 10 treatments over 10-20 days (Monday-Friday) in the absence of disease progression or unacceptable toxicity. Patients undergo magnetic resonance imaging (MRI) during screening and follow-up and undergo collection of blood samples throughout the trial. Patients also undergo lumbar puncture LP or Ommaya reservoir tap for cerebrospinal fluid (CSF) sample collection during screening and follow-up.

After completion of study treatment, patients are followed up at 1 month and then every 3 months for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative

  * Assent, when appropriate, will be obtained per institutional guidelines
* ≥ 18 years
* Karnofsky performance status (KPS) ≥ 60
* Ability to read and understand English or Spanish for questionnaires, or ability to complete questionnaires using certified interpreter
* Histologically confirmed breast cancer or non-small cell lung cancer
* Leptomeningeal disease established either radiographically and/or CSF cytology
* Absolute neutrophil count (ANC) ≥ 1,000/mm^3
* Hemoglobin ≥ 8 g/dL
* Platelet ≥ 100,000/mm^3
* Creatinine clearance of ≥ 50 mL/min per 24 hour urine test or the Cockcroft-Gault formula
* Women of childbearing potential (WOCBP): negative urine or serum pregnancy test

  * If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Agreement by females and males of childbearing potential to use an effective method of birth control or abstain from heterosexual activity for the course of the study through at least 1 month after the last dose of protocol therapy

  * Childbearing potential defined as not being surgically sterilized (men and women) or have not been free from menses for > 1 year (women only)

Exclusion Criteria:

* Chemotherapy, biological therapy, immunotherapy within 7 days prior to day 1 of protocol therapy
* Any prior radiation that in the opinion of the investigator unable to respect normal tissue tolerances and preclude craniospinal irradiation
* Patients with multiple or serious major neurologic symptoms (including encephalopathy) per physician / investigator assessment
* Patients with extensive, uncontrolled extracranial systemic disease
* Patients without reasonable systemic treatment options per physician / investigator
* Other clinically significant uncontrolled illness per opinion of physician / investigator
* Patients with a history or evidence of HIV infection (unless on effective anti-retroviral therapy with undetectable viral load based on prior tests within 6 months are eligible for this trial)
* Patients with history or evidence of chronic hepatitis B virus (HBV) infection (unless HBV viral load is undetectable based on prior tests and on suppressive therapy)
* Patients with a history or evidence of hepatitis C virus (HCV) infection unless treated and cured. (Patients with HCV infection who are currently on treatment are eligible if they have an undetectable HCV viral load based on prior tests)
* Other active malignancy. Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the study are eligible for this trial
* Females only: Pregnant or breastfeeding
* Any other condition that would, in the investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures
* Unable to undergo MRI brain and spine with gadolinium contrast
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-05-05 (Actual); Primary Completion 2028-10-02 (Estimated); Study Completion 2028-10-02 (Estimated)

PRIMARY OUTCOMES:
Central nervous system (CNS)-progression free survival | From start of treatment to CNS relapse, CNS progression, death (from any cause), or last contact, whichever occurs first, assessed up to 1 year
  Will be estimated using the Kaplan-Meier estimator, and its associating 95% confidence limit will be calculated using the logit transformation and the Greenwood variance estimate.

SECONDARY OUTCOMES:
Radiographic response | Every 3 months after treatment until CNS disease progression or death, assessed up to 1 year
  Will be assessed per European Organization for Research and Treatment of Cancer (EORTC) Response Assessment in Neuro-Oncology. Will be characterized using a (generalized) linear mixed effects model.
Quality of life | At baseline, 1 month, and every 3 months until CNS disease progression or death, assessed up to 1 year
  Will be assessed per EORTC Quality-of-Life Questionnaire Brain 20, EORTC Core Quality-of-Life Questionnaire 30, Patient Reported Outcome Measurement Information System (PROMIS) Anxiety short form and PROMIS Cognition short form. Will be characterized using a (generalized) linear mixed effects model.
Incidence of adverse events | Up to 30 days after the last day of treatment
  Will be assessed and graded according to the Common Terminology Criteria for Adverse Events version 5.0. Will be tabulated to show the number and percentage as well as the timing, severity, and attribution of the toxicity.
Overall survival | From start of treatment to death (from any cause), or last contact, whichever occurs first, assessed up to 1 year
  Will be estimated using the Kaplan-Meier estimator, and its associating 95% confidence limit will be calculated using the logit transformation and the Greenwood variance estimate.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie M Yoon, Principal Investigator — City of Hope Medical Center
Locations (2):
- United States (2):
  - City of Hope Medical Center, Duarte, California
  - City of Hope at Irvine Lennar, Irvine, California